CLINICAL TRIAL: NCT02839837
Title: The Benefits of Acute Aerobic Exercise on Neuroplastic Potential in Depression
Brief Title: Acute Aerobic Exercise and Neuroplasticity in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro#00050872
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Depression; Depressive Disorder
Keywords: Depression; Depressive Disorder; Exercise; Neuroplasticity; Non-invasive brain stimulation; Healthy Control
MeSH Terms: conditions — Depression; Depressive Disorder; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Depressed and non-depressed controls (Experimental): All participants will participate in three different conditions: Low intensity aerobic exercise and paired associative stimulation, high intensity aerobic exercise and paired associative stimulation, no exercise control and paired associative stimulation. The order of conditions will be randomized.
  Interventions: Behavioral: Aerobic Exercise; Device: Paired Associative Stimulation

INTERVENTIONS:
Behavioral: Aerobic Exercise — Aerobic exercise will be performed on a stationary cycle ergometer for 15 minutes at an intensity of 35% heart rate reserve or 70% heart rate reserve. During the control condition the participant will remain seated on the stationary cycle for 15 minutes and will not perform exercise.
Device: Paired Associative Stimulation — After aerobic exercise participants will receive a paired associative stimulation (PAS) paradigm. PAS consists of paired brain and peripheral nerve stimuli. Participants will receive 200 paired stimuli. Peripheral nerve stimulation will be delivered to the median nerve at the level of the wrist via electrical stimulation at 300% perceptual threshold. Brain stimulation will be delivered via transcranial magnetic stimulation (TMS) over the hand knob of the motor cortex at an intensity that elicits a 1mV response in the contralateral abductor pollicis brevis muscle. During each paired stimulation, peripheral nerve stimulation will precede the TMS stimulation by 25ms.

SUMMARY:
Depression is associated with a disruption in the mechanisms that regulate neuroplasticity. Effective treatment and rehabilitation of depression, and other neurological and neuropsychiatric disorders, relies on neuroplasticity. Thus, identifying therapies that enhance neuroplasticity (neuroplastic adaptation) are vital in the comprehensive treatment of depression. Aerobic exercise training has been demonstrated to have antidepressant properties and single bouts of aerobic exercise may provide short-term improvements in affective states in depression. Furthermore, acute aerobic exercise may enhance the response to known neuroplasticity-inducing paradigms. However, it is unclear if aerobic exercise can influence neuroplasticity in depression and the neurobiological mechanisms underlying acute neuroplastic changes are not well understood in depressed and healthy cohorts. Thus, the purpose of this project is to examine the acute effects of aerobic exercise on neuroplastic, neurobiological, and mood indices of depression.

DETAILED DESCRIPTION:
The investigators will determine the effects of exercising at two different intensities (compared to a control non-exercise condition) on neuroplastic potential in depressed and non-depressed subjects. To accomplish this aim, the investigators will have subjects ride a cycle ergometer at intensities set to elicit 35% (low) and 70% (high) of heart rate reserve (((220 - age) - resting heart rate) x 35% or 70%) + resting heart rate). Prior to, and immediately after exercise participants will have their neuroplastic potential tested via transcranial magnetic stimulation (TMS), blood specimens sampled, and mood changes assessed (methods detailed below). These assessments will occur at these time points and then every 15 minutes for 1 hour after exercise.

Neuroplastic potential will be assessed using TMS. TMS-induced motor evoked potentials (MEP's) will be recorded from the abductor pollicis brevis as a way to measure changes in the excitability of the corticospinal tract in response to exercise and paired associative stimulation. Serum brain-derived neurotrophic factor (BDNF) and cortisol levels will be obtained through blood specimen samples in order to examine the potential exercise-induced changes in known stress- and neuroplasticity-related biomarkers. Mood and affect will be surveyed using the Activation-Deactivation Checklist (AD ACL), feeling scale (FS), and felt arousal scale (FAS). These measures will permit the assessment of exercise-induced changes in mood and affect.

ELIGIBILITY:
Inclusion Criteria:

For all:

1. age 18-50 year old.
2. ability to provide informed consent.

Further inclusion criteria for participants with depression:

1. meets criteria for unipolar depression assessed using the Mini-international Neuropsychiatric Interview (MINI)
2. a Montgomery Asberg Depression Rating Scale (MADRS) score of 20 or greater
3. current depressive episode began no longer than 3 years earlier
4. psychoactive drug free or have maintained a stable dose of up to one antidepressant medication for four weeks prior to study participation

Further inclusion criteria for control participants:

1. does not meet criteria for unipolar depression assessed using the MINI
2. a MADRS score of 6 or less
3. no history or previous diagnosis of depression

Exclusion Criteria (for all participants):

* primary diagnosis of another Axis 1 disorder
* secondary diagnosis of a psychotic disorder, cognitive disorder, substance-related disorder, or obsessive compulsive disorder
* illicit drug use or alcohol abuse
* current smoker
* history of seizures
* other diagnosed neurological or musculoskeletal disorder/injury, uncontrolled cardiovascular or metabolic disease
* resting blood pressure > 200mmHg systolic or 100mmHg diastolic
* electronic or metal implants
* current participation in a structured exercise program
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in peak to peak MEP amplitude (mV) | From baseline to one hour post-PAS

SECONDARY OUTCOMES:
Change in serum BDNF (ng/ml) | From baseline to one hour post-exercise
Change in serum cortisol (ng/ml) | From baseline to one hour post-exercise

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gregory, P.T., Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Stroke Recovery Research Center, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No